CLINICAL TRIAL: NCT05300529
Title: Effectiveness of Vestibular Rehabilitation for Improving Health Status in Patients With Fibromyalgia. Randomized Clinical Trial
Brief Title: Effectiveness of Vestibular Rehabilitation for Improving Health Status in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Ana Peinado Rubia, PhD student, principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UjaFM
Record Dates: First submitted 2022-01-24; First posted 2022-03-29 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Fibromyalgia; Vestibular Disease; Postural Balance; Vestibular Rehabilitation
Keywords: Fibromyalgia; Vestibular Disease; Postural Balance; Vestibular Rehabilitation
MeSH Terms: conditions — Fibromyalgia; Vestibular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Rehabilitation Exercises (Experimental): Vestibular Rehabilitation Exercises focused on eye stabilization and Vestibulo-Oculo Reflex (VOR). Two sessions/week supervised by researcher (40 min) and conducting exercises at home 2 times/day, 5 days/week. (15-20 min)
  Interventions: Other: Vestibular Rehabilitation Exercises
- Conventional Rehabilitation exercises (Sham Comparator): Conventional rehabilitation exercises: stretching and walking. Two sessions/week supervised by researcher (40 min) and conducting exercises at home 2 times/day, 5 days/week. (15-20 min)
  Interventions: Other: Conventional Rehabilitation exercises

INTERVENTIONS:
Other: Vestibular Rehabilitation Exercises — The Vestibular Rehabilitation program focuses on stabilizing the gaze and gaining the Vestibular Ocular Reflex (VOR). The general mechanisms of recovery from vestibular injuries are vestibular adaptation and replacement exercises, which are designed to improve gaze stability and the interaction between sight and the vestibular system during head movements. The exercises will be carried out progressively according to the tolerance of the patient, varying the stimulus in intensity and frequency.
  Arms: Vestibular Rehabilitation Exercises
Other: Conventional Rehabilitation exercises — The conventional rehabilitation program in which exercises are performed to improve joint range, flexibility, and gait. It will always be done with the eyes open, on a firm surface and will not include training in sensory strategies
  Arms: Conventional Rehabilitation exercises

SUMMARY:
The purpose of this study is to analyze the effectiveness of Vestibular Rehabilitation for improving balance and quality of life of patients with Fibromyalgia Syndrome (SFM). Recruited subjects will be randomly assigned to an experimental group or control group (placebo). The experimental group will receive a standard Vestibular Rehabilitation program focused on eye stabilization and Vestibulo-Ocular Reflex (VOR) gain with the aim of improving motor and sensory strategies, while the control group will carry out a conventional rehabilitation program that will not include sensory strategy training. The frequency of treatment for both groups will be twice/week, along with daily performing (2 times/day, 5 days/week) of exercises at home. The total duration will be 8 weeks. The outcome measure are: disease impact (FIQ), perceived vertigo (DHI), and confidence in balance (ABC), at pre-treatment, post-treatment, one month follow-up and three months follow-up.

DETAILED DESCRIPTION:
Fibromyalgia Syndrome (SFM) affects approximately 0.5 - 5% of the global population with ambiguity in diagnosis, physiopathology uncertainty and complex treatment.

Recent studies have shown frequent episodes of postural instability in SFM patients. This balance affectation seems to correlate with disturbances of quality of life, pain, impact of the disease, daily life activities and increased risk of falls. However, there is still controversy over the exact mechanism that explains this nonspecific balance disorder. Despite this preliminary finding of a possible visual and vestibular disorder, there are not known studies justifying the alteration of vestibular functions present in Fibromyalgia. Also, the are not certainty that Vestibular Rehabilitation (VR) provides short- and medium-term benefits.

Derived from the deficiencies observed in the revised literature, we propose to analyze the effectiveness of a Vestibular Rehabilitation program improving the balance and quality of life of people with Fibromyalgia Syndrome (SFM).

Therefore, a randomized, simple blind, two-group parallel controlled clinical trial has been designed to assess the effectiveness of Vestibular Rehabilitation treatment focused on eye stabilization exercises.

Subjects will be recruited from the Jaén Fibromyalgia Association (AFIXA) and randomly assigned to an experimental group or control group (placebo). Subjects who are diagnosed with SFM and between 18 and 70 years of age will be selected.

The experimental group will receive a standard Vestibular Rehabilitation program focused on the stabilization of the eye and gain of the Vestibulo-Oculo Reflex (VOR), while in the control group a conventional rehabilitation program will be carried out without visual stimulation. The frequency of treatment for both groups will be twice/week, along with daily exercises at home (2 times/day). The total duration will be 8 weeks. Measurements will be made in pretreatment, aftertreatment and one month follow-up and three months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years,
* Diagnostic for fibromyalgia as described by the 2016 American College of Rheumatology (ACR)

Exclusion Criteria:

* Cognitive impairment impacting ability to fill out the scales and questionnaires.
* Musculoskeletal surgical intervention in the preceding 6 months and/or acute traumatic pathology to the inferior limb(s).
* Musculoskeletal disease with deformity of the inferior limbs.
* Diagnosed with vestibular, visual and/or auditory pathology.
* Neurologic illness that could be the cause of a balance disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
FIQ (Fibromyalgia Impact Questionnaire) | Baseline
  Evaluates the impact of fibromyalgia on the patient's quality of life.The total score of the FIQ is from 0 to 100. A higher score means a greater impact of the disease on the patient.
FIQ (Fibromyalgia Impact Questionnaire) | at eight weeks
  Evaluates the impact of fibromyalgia on the patient's quality of life.The total score of the FIQ is from 0 to 100. A higher score means a greater impact of the disease on the patient.
FIQ (Fibromyalgia Impact Questionnaire) | at twelve weeks
  Evaluates the impact of fibromyalgia on the patient's quality of life.The total score of the FIQ is from 0 to 100. A higher score means a greater impact of the disease on the patient.
ABC-16 (Activities-specific Balance Confidence scale-16 items) | Baseline
  Evaluates the balance confidence in performing activities of daily living. The total score of the ABC-16 is from 0% to 100%, with higher values associated with higher balance confidence.
ABC-16 (Activities-specific Balance Confidence scale-16 items) | at eight weeks
  Evaluates the balance confidence in performing activities of daily living. The total score of the ABC-16 is from 0% to 100%, with higher values associated with higher balance confidence.
ABC-16 (Activities-specific Balance Confidence scale-16 items) | at twelve weeks
  Evaluates the balance confidence in performing activities of daily living. The total score of the ABC-16 is from 0% to 100%, with higher values associated with higher balance confidence.
DHI (Dizziness Handicap Inventory) | Baseline
  Evaluates the level of disability related to the impact of dizziness on daily function and quality of life. The total score of the DHI is from 0 to100 points. A higher score indicates a greater degree of disability due to the vertiginous symptoms.
DHI (Dizziness Handicap Inventory) | at eight weeks
  Evaluates the level of disability related to the impact of dizziness on daily function and quality of life. The total score of the DHI is from 0 to100 points. A higher score indicates a greater degree of disability due to the vertiginous symptoms.
DHI (Dizziness Handicap Inventory) | at twelve weeks.
  Evaluates the level of disability related to the impact of dizziness on daily function and quality of life. The total score of the DHI is from 0 to100 points. A higher score indicates a greater degree of disability due to the vertiginous symptoms.

SECONDARY OUTCOMES:
CSI (Central Sensitization Inventory) | Baseline
  Evaluates a wide range of somatic and emotional symptoms common to central sensitization syndromes (CSS). The total score of the CSI from 0 to 100. Higher scores indicate greater severity of symptoms.
CSI (Central Sensitization Inventory) | at eight weeks
  Evaluates a wide range of somatic and emotional symptoms common to central sensitization syndromes (CSS). The total score of the CSI from 0 to 100. Higher scores indicate greater severity of symptoms.
CSI (Central Sensitization Inventory) | at twelve weeks.
  Evaluates a wide range of somatic and emotional symptoms common to central sensitization syndromes (CSS). The total score of the CSI from 0 to 100. Higher scores indicate greater severity of symptoms.
PCS (Pain Catastrophizing Scale) | Baseline
  Evaluates the patient's catastrophic thoughts. The total score of the PCS from 0 to 52. Higher scores indicate a greater presence of catastrophic thoughts.
PCS (Pain Catastrophizing Scale) | at eight weeks
  Evaluates the patient's catastrophic thoughts. The total score of the PCS from 0 to 52. Higher scores indicate a greater presence of catastrophic thoughts.
PCS (Pain Catastrophizing Scale) | at twelve weeks.
  Evaluates the patient's catastrophic thoughts. The total score of the PCS from 0 to 52. Higher scores indicate a greater presence of catastrophic thoughts.
TSK (Tampa Scale for Kinesiophobia) | Baseline
  Evaluates fear of movement to injury. The total score of the TSK from 11 to 44 points. Higher scores indicate a greater fear of movement.
TSK (Tampa Scale for Kinesiophobia) | at eight weeks
  Evaluates fear of movement to injury. The total score of the TSK from 11 to 44 points. Higher scores indicate a greater fear of movement.
TSK (Tampa Scale for Kinesiophobia) | at twelve weeks.
  Evaluates fear of movement to injury. The total score of the TSK from 11 to 44 points. Higher scores indicate a greater fear of movement.
VAS-pain (Visual Analogue Scale) | Baseline
  Evaluates the pain on a numerical scale from 0 to 10. Higher scores indicate more pain
VAS-pain (Visual Analogue Scale) | at eight weeks
  Evaluates the pain on a numerical scale from 0 to 10. Higher scores indicate more pain
VAS-pain (Visual Analogue Scale) | at twelve weeks
  Evaluates the pain on a numerical scale from 0 to 10. Higher scores indicate more pain
SF-12 (12-Item Short Form Survey) | Baseline
  Evaluates the impact of health on an individual's everyday life. Used as a quality of life measure.
SF-12 (12-Item Short Form Survey) | at eight weeks
  Evaluates the impact of health on an individual's everyday life. Used as a quality of life measure.
SF-12 (12-Item Short Form Survey) | at twelve weeks
  Evaluates the impact of health on an individual's everyday life. Used as a quality of life measure.
FES-I (Falls Efficacy Scale-International) | Baseline
  Evaluates the fear of falling. The total score of the FES-I from 16 to 64 points. Higher scores indicate greater fear of falling.
FES-I (Falls Efficacy Scale-International) | at eight weeks
  Evaluates the fear of falling. The total score of the FES-I from 16 to 64 points. Higher scores indicate greater fear of falling.
FES-I (Falls Efficacy Scale-International) | at twelve weeks
  Evaluates the fear of falling. The total score of the FES-I from 16 to 64 points. Higher scores indicate greater fear of falling.
FSS (Fatigue Severity Scale) | Baseline
  Evaluates severity of fatigue. Higher scores indicate a greater severity of fatigue
FSS (Fatigue Severity Scale) | at eight weeks
  Evaluates severity of fatigue. Higher scores indicate a greater severity of fatigue
FSS (Fatigue Severity Scale) | at twelve weeks
  Evaluates severity of fatigue. Higher scores indicate a greater severity of fatigue
20-item JAEN screening tool | Baseline
  Evaluates balance and neuromotor function in patients with fibromyalgia. Thd total scale of the Jaen-Screening Tools, from 0 to 80 points. A higher score indicates a greater degree of balance disorder.
20-item JAEN screening tool | at eight weeks
  Evaluates balance and neuromotor function in patients with fibromyalgia. Thd total scale of the Jaen-Screening Tools, from 0 to 80 points. A higher score indicates a greater degree of balance disorder.
20-item JAEN screening tool | at twelve weeks
  Evaluates balance and neuromotor function in patients with fibromyalgia. Thd total scale of the Jaen-Screening Tools, from 0 to 80 points. A higher score indicates a greater degree of balance disorder.
SVV (Subjective Visual Vertical) | baseline
  Evaluates the perception of verticality, measured using the Subjective Visual Vertical (SVV) test using a virtual reality device.
SVV (Subjective Visual Vertical) | at eight weeks
  Evaluates the perception of verticality, measured using the Subjective Visual Vertical (SVV) test using a virtual reality device.
SVV (Subjective Visual Vertical) | at twelve weeks
  Evaluates the perception of verticality, measured using the Subjective Visual Vertical (SVV) test using a virtual reality device.
Stabilometric Platform | Baseline
  Instrument composed of resistive pressure sensors, used to measure the static or postural balance. The test was performed under both eyes-open and eyes-closed conditions.
Stabilometric Platform | at eight weeks
  Instrument composed of resistive pressure sensors, used to measure the static or postural balance. The test was performed under both eyes-open and eyes-closed conditions.
Stabilometric Platform | at twelve weeks
  Instrument composed of resistive pressure sensors, used to measure the static or postural balance. The test was performed under both eyes-open and eyes-closed conditions.
Therapeutic Adherence at home | Throughout the intervention phase, eight weeks
  It assesses adherence to home treatment through a weekly record diary, where patients must record the number of times a day they perform the prescribed exercises, with a range of 0 to 80. Higher scores indicate greater adherence to home treatment. A score of 80 indicates 100% adherence.
Satisfaction level | at eight weeks
  Evaluates the level of satisfaction using a Likert scale, with five response options, from "very dissatisfied" to "very satisfied". The total score of 0-24. A high score indicates greater satisfaction
GRC (Global Change Rating Scales) | at eight weeks
  Assesses whether the patient's health status has improved or deteriorated after the treatment received, with ten response options ranging from "the worst it could be" to "the best it could be"

OTHER OUTCOMES:
Height (Anthropometrics Data) | Baseline
  Patient height measured in meters (m)
Weight (Anthropometrics Data) | Baseline
  Patient's body weight in kilograms (kg)
Body Mass Index (Anthropometrics Data) | Baseline
  Weight and height will be combined to report body mass index in kg/m^2
Demographics Data | Baseline
  Registration of information provided by the patient on sex, age, education level. occupation and civil status

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Lomas-Vega, PhD, Principal Investigator — University of Jaén
Locations (1):
- University os Jaén, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No